CLINICAL TRIAL: NCT04816019
Title: A Phase I Study to Determine Safety, Tolerability and Immunogenicity of Intranasal Administration of the COVID Vaccine ChAdOx1 nCOV-19 in Healthy UK Adults
Brief Title: A Study of Intranasal ChAdOx1 nCOV-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: COV008
Record Dates: First submitted 2021-03-15; First posted 2021-03-25 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus
Keywords: Covid-19; ChAdOx1 nCov19; SARS-CoV-2; Vaccine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1a: Low Dose (Experimental): A single, Covid-19 vaccine naive volunteer will receive a single dose of 5x10^9vp ChAdOx1 nCOV-19 IN.
  Volunteers in Group 1a & b will be randomized to receive booster dose of 5 x 10^9vp ChAdOx1 IN or no booster
  Interventions: Biological: ChAdOx1 nCov-19
- Group 1b: Low dose (Experimental): 5 Covid-19 vaccine naive volunteers will receive a single dose of 5x10^9vp ChAdOx1 nCOV-19 IN.
  Volunteers in Group 1a & b will be randomized to receive booster dose of 5 x 10^9vp ChAdOx1 IN or no booster
  Interventions: Biological: ChAdOx1 nCov-19
- Group 2a: High Dose (Experimental): 3 Covid-19 vaccine naivevolunteers will receive a single dose of 5x10^10vp ChAdOx1 nCOV-19 IN.
  Volunteers in Group 2a & b will be randomized to receive booster dose of 5 x 10^10vp ChAdOx1 IN or no booster
  Interventions: Biological: ChAdOx1 nCov-19
- Group 2b: High Dose (Experimental): Up to 15 Covid-19 vaccine naive volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCOV-19 IN.
  Volunteers in Group 2a & b will be randomized to receive booster dose of 5 x 10^10vp ChAdOx1 IN or no booster
  Interventions: Biological: ChAdOx1 nCov-19
- Group 3: Intermediate Dose (Experimental): Up to 18 Covid-19 vaccine naive volunteers will receive a single dose of 2x10^10vp ChAdOx1 nCOV-19 IN.
  Volunteers will be randomized to receive booster dose of 2 x 10^10vp ChAdOx1 IN or no booster
  Interventions: Biological: ChAdOx1 nCov-19
- Group 4: High Dose, vaccinated boost (Experimental): 6 volunteers, previously vaccinated with two doses of ChAdOx1 nCoV-19 IM will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 IN.
  Interventions: Biological: ChAdOx1 nCov-19
- Group 5: High Dose, vaccinated boost (Experimental): 6 volunteers, previously vaccinated with two doses of BNT162b IM will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 IN.
  Interventions: Biological: ChAdOx1 nCov-19

INTERVENTIONS:
Biological: ChAdOx1 nCov-19 — A single dose of ChAdOx1 nCov-19 delivered intranasally (IN)

SUMMARY:
Open label, dose escalation study to investigate:

1. Safety, tolerability and immunogenicity of one or two doses of intranasal ChAdOx1 nCOV-19, in vaccine naïve individuals, with randomisation between one and two dose groups.
2. Safety, tolerability and immunogenicity of intranasal ChAdOx1 nCOV-19, given as a booster dose in individuals who have had two intramuscular COVID-19 vaccinations.

DETAILED DESCRIPTION:
The study will include up to 54 healthy adult participants, divided into five groups. Groups 1-3 will consist of vaccine-naïve volunteers and groups 4-5 will consist of volunteers who have received 2 doses of IM COVID-19 vaccine.

Groups 1-3 will receive three vaccine dose levels (low i.e. 5x10^9vp, high i.e. 5x10^10 VP, and moderate i.e. 2x10^10 VP ChAdOx1 nCOV-19 IN). The low and high dose groups will each have safety lead-in subgroups. All volunteers will be consented for receipt of a booster vaccine at approximately 4 weeks post first vaccine. All volunteers will be randomly allocated 1:1 to receive an intranasal booster vaccine as indicated, stratified by first dose level.

Group 4 will consist of volunteers who have received 2 intramuscular doses of ChAdOx1 nCoV-19, at least eight weeks apart, and group 5 will consist of volunteers who have received 2 intramuscular doses of BNT162b, at least three weeks apart. Both of these groups will receive a single standard dose (5x1010vp) on intranasal ChAdOx1 nCOV-19.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1, 2 and 3 only: Healthy adults aged 18-55 years (Note, prior to implementation of SA001, a single participant under the age of 30 was enrolled in group 1a. This participant will be retained for follow-up but will not receive a booster vaccine, in light of the new age restrictions. Between the implementation of SA001 and implementation of SA003, only those aged 30-40 years were eligible.
* Groups 4 and 5 only: Healthy adults aged 30-55 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner and access all medical records when relevant to study procedures.
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of screening and vaccination.
* Agreement to refrain from blood donation during the course of the study.
* Provide written informed consent.
* Group 4 only: Prior receipt of 2 doses of ChAdOx1 nCoV-19 intramuscularly, with an interval of at least 8 weeks between the intramuscular doses, and with the second dose a minimum of 12 weeks prior to enrolment
* Group 5 only: Prior receipt of 2 doses of BNT162b2 intramuscularly, with an interval of at least 3 weeks between the intramuscular doses, and with the second dose a minimum of 12 weeks prior to enrolment

Acceptable forms of contraception for female volunteers include:

* Established use of oral, injected or implanted hormonal methods of contraception.
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Total abdominal hysterectomy.
* Bilateral tubal Occlusion Barrier methods of contraception (condom or occlusive cap with spermicide).
* Male sterilisation, if the vasectomised partner is the sole partner for the subject.
* True abstinence, when this is in line with the preferred and usual lifestyle of the subject.
* Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to IMP, and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* Receipt or planned receipt of any vaccine other than the study intervention within 28 days before and after each study vaccination.
* Participation in COVID-19 prophylactic drug trials for the duration of the study. (Note: Participation in COVID-19 treatment trials is allowed in the event of hospitalisation due to COVID-19. The study team should be informed as soon as possible.)
* Groups 1, 2 and 3 only: Prior receipt of an investigational or licensed vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus vaccines).
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months, except topical steroids or short-term oral steroids (course lasting <14 days).
* Any autoimmune conditions, except mild psoriasis, well-controlled autoimmune thyroid disease, vitiligo or stable coeliac disease not requiring immunosuppressive or immunomodulatory therapy.
* History of allergic disease or reactions likely to be exacerbated by any component of ChAdOx1 nCoV-19.
* Any history of angioedema.
* Any history of anaphylaxis.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of any organic central nervous system disorder or any functional disorder involving neurological symptoms
* History of serious psychiatric condition likely to affect participation in the study (e.g. ongoing severe depression, history of admission to an in-patient psychiatric facility, recent suicidal ideation, history of suicide attempt, bipolar disorder, personality disorder, alcohol and drug dependency, severe eating disorder, psychosis, use of mood stabilisers or antipsychotic medication).
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture, or continuous anticoagulation e.g. with warfarin
* History of confirmed major thrombotic event (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism), or
* History of antiphospholipid syndrome
* Prior receipt of unfractionated heparin
* History of heparin induced thrombocytopenia
* Any other serious chronic illness requiring hospital specialist supervision.
* Chronic respiratory diseases, including mild asthma (resolved childhood asthma is allowed).
* Chronic cardiovascular disease (including hypertension), gastrointestinal disease, liver disease (except Gilberts Syndrome), renal disease, endocrine disorder (including diabetes) and neurological illness (excluding migraine).
* Nasal pathology (e.g. congenital abnormalities such as an abnormal septum or polyps, previous cauterisation, rhinoplasty or nasal surgery of any kind, recurrent epistaxis).
* Seriously overweight (BMI≥40 Kg/m2) or underweight (BMI≤18 Kg/m2).
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Any clinically significant abnormal finding on screening biochemistry, haematology blood tests or urinalysis.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Groups 1, 2 and 3 only: Living in the same household as any vulnerable groups at risk of severe COVID-19 disease (as per PHE guidance).
* Groups 1, 2 and 3 only: Membership of any group identified by JCVI at the time of enrolment as being eligible for priority vaccination (i.e. ahead of the typical member of the individual's age cohort).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of intranasal administration of ChAdOx1 nCov-19 in healthy adult volunteers: Occurrence of solicited signs and symptoms | 7 days
  Occurrence of solicited local and systemic reactogenicity signs and symptoms for 7 days following vaccination
Investigate the safety and tolerability of intranasal administration of ChAdOx1 nCov-19 in healthy adult volunteers: Occurrence of unsolicited signs and symptoms | 28 days
  Occurrence of unsolicited adverse events (AEs) for 28 days following vaccination
Investigate the safety and tolerability of intranasal administration of ChAdOx1 nCov-19 in healthy adult volunteers: Occurrence of adverse events as identified by change in baseline safety laboratory measures | 7 or 35 days
  Change from baseline for safety laboratory measures (hematology and biochemistry) at Day 7 (and Day 35 for 2 dose groups only).
  Safety laboratory measures include clinical blood tests for full blood count, liver function and renal function as graded on a predetermined toxicity grading scale.
Investigate the safety and tolerability of intranasal administration of ChAdOx1 nCov-19 in healthy adult volunteers: Occurrence of serious adverse events (SAEs) | 4 months
  Occurrence of SAEs and AWESIs collected throughout the trial

SECONDARY OUTCOMES:
Assess the mucosal immune response to intranasal administration of one or two doses of ChAdOx1 nCov-19 in healthy adult volunteers | 112 days
  Quantification of spike-binding mucosal antibody, collected using SAM strips at D0, D7, D14, D28, D42 (2 dose groups only), D56, D112.
  Includes characterisation of dose-response relationship

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Douglas, Dr, Principal Investigator — University of Oxford
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Nakahashi-Ouchida R, Fujihashi K, Kurashima Y, Yuki Y, Kiyono H. Nasal vaccines: solutions for respiratory infectious diseases. Trends Mol Med. 2023 Feb;29(2):124-140. doi: 10.1016/j.molmed.2022.10.009. Epub 2022 Nov 23. PMID 36435633